CLINICAL TRIAL: NCT01910740
Title: Optimising Rehabilitation Outcomes in Frail Older Adults: Effects of Increasing the Amount of Physical Activity
Brief Title: Mobility in Older People
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: La Trobe University (Other)
Collaborators: Austin Health (Other Government)
Responsible Party: Principal Investigator, Meg Morris, Professor Meg Morris, La Trobe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHMRC - 1042680
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Frail Older People Undergoing Inpatient Rehabilitation
Keywords: Randomized Controlled Trial; Exercise Movement Techniques; Frail Elderly; Gait
MeSH Terms: interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Physical Activity (Experimental): Participants in the Enhanced Physical Activity group will receive a program of enhanced physical activity in addition to the usual care.
  Interventions: Other: Enhanced Physical Activity; Other: Usual Care
- Usual Care (Active Comparator): The Usual Care group will receive usual therapy provided by a multidisciplinary team and social interaction.
  Interventions: Other: Usual Care; Other: Social Interaction

INTERVENTIONS:
Other: Enhanced Physical Activity — Individually tailored programs focused on increasing the amount of time participants spend performing mobility activities, particularly standing and walking in the late afternoons and evenings and on weekends. These participants will be provided with one or two extra sessions on weekdays and two extra sessions on weekend days for the duration of their rehabilitation stay.
  Arms: Enhanced Physical Activity
Other: Usual Care — Therapy provided by a multidisciplinary team which includes physiotherapy and occupational therapy on weekdays with other allied health input (eg speech pathology, social work) as indicated. Medical and nursing care is also provided seven days a week.
Other: Social Interaction — To control for the extra hours of physical activity that the experimental group receives, participants in the control group shall have additional activities such as card and board games, conversation or reading as well as upper limb exercises and other physical activities that have minimal impact on ambulant mobility.
  Arms: Usual Care

SUMMARY:
The main aim of this study is to investigate whether increasing the amount of physical activity in frail older people during hospital based rehabilitation is associated with better mobility outcomes compared to usual care. A second aim is to investigate whether this physical activity intervention is associated with improvements in health related quality of life. Finally we plan to investigate whether increasing the amount of physical activity during rehabilitation is cost effective, measured from a health system perspective, compared with usual care.

Older people receiving inpatient rehabilitation will be randomly assigned to an intervention group, who will receive extra physical activity on weekdays and weekends or a control group, who will receive additional activities based on social interaction. The activity sessions will be individualized to the particular participant. Both groups of people will be assessed at baseline, discharge from hospital and at 6 months following discharge. The intervention group will be provided with one or two extra sessions on weekdays and two extra sessions on weekends for the duration of their rehabilitation stay. To account for the extra physiotherapy time that the intervention group receives, the people in the control group will spend the same amount of time performing other activities, such as cards, board games or reading, whilst seated. To ensure the safety of the participants in this study, each physical activity session will be supervised by either a physiotherapist or allied health assistant.

Hypothesis 1: The primary hypothesis is that, compared with usual care, increasing the amount of physical activity in frail older people during rehabilitation will lead to more optimal mobility at discharge, as measured by gait speed.

Secondary hypotheses are that, compared with usual care, increasing the amount of physical activity during rehabilitation will:

Hypothesis 2: lead to significantly greater improvements in mobility and function both at discharge and six months following discharge.

Hypothesis 3: lead to better quality of life six months following hospital discharge, measured using the EuroQol Health (EQ5D) Questionnaire and the EuroQol-Visual Analogue Scale (EQ-VAS).

Hypothesis 4: be cost effective compared to usual care

ELIGIBILITY:
Inclusion Criteria:

* over 60 years of age
* a goal of admission is to 'improve weight-bearing mobility or improve walking' as determined by either the admission referral or the treating therapist

Exclusion Criteria:

* specific medical restrictions that limit mobilisation (e.g. non weight bearing)
* if already enrolled in a different Randomised Controlled Trial
* previously enrolled in the current trial
* the primary reason for admission is awaiting a residential care placement
* the primary reason for admission is for carer training

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Gait Velocity | Discharge (Average Duration of Hospital Stay is 3 weeks)
  Gait velocity will be measured using the 6 metre walk test

SECONDARY OUTCOMES:
Gait Velocity | 6 Months Follow Up (post discharge)
  Gait velocity will be measured using the 6 metre walk test

CONTACTS AND LOCATIONS:
Overall Officials: Meg Morris, PhD, Principal Investigator — La Trobe University
Locations (1):
- Heidelberg Repatriation Hospital, Austin Health, Heidelberg, Victoria, Australia

REFERENCES:
- [Derived] Said CM, McGinley JL, Szoeke C, Workman B, Hill KD, Wittwer JE, Woodward M, Liew D, Churilov L, Bernhardt J, Morris ME. Factors associated with improved walking in older people during hospital rehabilitation: secondary analysis of a randomized controlled trial. BMC Geriatr. 2021 Jan 31;21(1):90. doi: 10.1186/s12877-021-02016-0. PMID 33517882
- [Derived] Said CM, Morris ME, McGinley JL, Szoeke C, Workman B, Liew D, Hill K, Woodward M, Wittwer JE, Churilov L, Ventura C, Bernhardt J. Evaluating the effects of increasing physical activity to optimize rehabilitation outcomes in hospitalized older adults (MOVE Trial): study protocol for a randomized controlled trial. Trials. 2015 Jan 15;16:13. doi: 10.1186/s13063-014-0531-y. PMID 25588907